CLINICAL TRIAL: NCT06455215
Title: The Community Garden Health Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: University of Hawaii Cancer Research Center (Other); Coalition for a Tobacco Free Arkansas (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 297248; OT2HL156812 (NIH)
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-07

CONDITIONS: Fruit and Vegetable Consumption
Keywords: food security, community gardens, fruit/vegetable consumption

STUDY DESIGN:
Intervention Model Description: Randomization will occur at the garden level. Four gardens will be randomized to the intervention and three gardens to the control group. The participants assigned to the four gardens in the intervention group will receive an 8-week intervention that includes 1) educational materials, 2) healthy cooking demonstrations, 3) food and transportation support and 4) garden social activities. The control garden group will not receive an intervention during this time period which allows us to evaluate differences in the primary and secondary outcomes in the intervention and control groups at 8 weeks and 6 months.
  The control group will receive the delayed 8-week intervention one month after the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Garden intervention (Experimental): The gardens in the intervention group will receive an 8-week intervention that includes 1) educational materials, 2) healthy cooking demonstrations, food and transportation support and 3) garden social activities.
  Interventions: Behavioral: Community garden activities
- Delayed intervention (Active Comparator): The control group will be asked to abstain from intervention activities during the 8 week period. The control group will receive the delayed 8-week intervention one month after the intervention group.
  Interventions: Behavioral: Community garden activities

INTERVENTIONS:
Behavioral: Community garden activities — The gardens in the intervention group will receive an 8-week intervention that includes 1) educational materials, 2) healthy cooking demonstrations, food and transportation support and 3) garden social activities. The control group will be asked to abstain from intervention activities. The control group will receive the delayed 8-week intervention one month after the intervention group.

SUMMARY:
The goals of this community-based clinical trial are to examine the association between community garden participation and 1) fruit and vegetable intake (primary outcome) and 2) access to healthy food (secondary outcome) among adults aged 18-95 living in low resource communities. Gardens will be randomized to the intervention (n=4 gardens) or control group (delayed intervention, n=3 gardens). Participants will be assigned to one of seven community gardens to receive an 8-week intervention. During the intervention, participants will be asked to volunteer in the garden, participate in garden social activities, participate in healthy cooking demonstrations and educational sessions. Participants will receive educational materials as well. To assess the effects of the intervention, participants will receive a baseline, 8-week, and 6-month survey. Outcome measures will be compared between the intervention and control groups.

DETAILED DESCRIPTION:
Food insecurity is a major cause of chronic diseases and is highest in the nation in Arkansas. Evidence shows that community gardens and healthy cooking demonstration can reduce food insecurity by 1) increasing access to healthy foods and 2) promoting healthy food consumption. Community garden participation is one factor that can influence healthy food consumption such as fruit and vegetable intake. The goals of this community-based clinical trial are to examine the association between community garden participation and 1) fruit and vegetable intake (primary outcome) and 2) access to healthy food (secondary outcome) among adults aged 18-95 living in low resource communities. Participants will be assigned to one of seven community gardens to receive an 8-week intervention. During the intervention participants will be asked to volunteer in the garden, participate in garden social activities, participate in healthy cooking demonstrations and educational sessions. Participants will receive educational materials as well. Four of the gardens will be randomized to the intervention group and three to the delayed intervention group. To assess the effects of the intervention, participants will receive a baseline, 8-week, and 6-month survey. Other measures that we will examine include food security; sociodemographics; physical activity; life satisfaction; perceived stress; neighborhood collective efficacy; self-efficacy; individual level social determinants of health; community engagement; and knowledge, attitudes, and satisfaction related to gardening and cooking.

ELIGIBILITY:
Inclusion Criteria:

1. Arkansas resident aged 18-95;
2. live in community within 1 mile radius of a participating garden;
3. speak English;
4. willingness to participate in the garden as a volunteer during the study intervention period;
5. not previously participated in the garden as a volunteer in past 6 months;
6. scores as food insecure on 1 of any of the food security measures (i.e. food did not last, could not eat balanced meal, cut the size or skip meals and frequency at which this happens, eat less than you think you should, were hungry but did not eat);
7. written informed consent;
8. working phone, home address, and email;

10) willingness to complete all survey assessments.

Exclusion Criteria:

* Does not live within 1 mile radius of a participating garden.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Fruit and vegetable intake | From baseline to 8 weeks (end of intervention) and 6-months post intervention
  We will use the five factor screener that is used to approximate intake of fruit juices, fruit, green leafy vegetables, other vegetables, tomato-based sauces, potatoes, and beans

SECONDARY OUTCOMES:
Access to healthy foods | From baseline to 8 weeks (end of intervention) and 6-months post intervention
  We will use the the Perceived Availability of the Healthy Food Scale. Participants will be asked to think of the neighborhood area (1 mile radius) and the extent to which they feel that the foods are of high quality, available, and are low fat.

CONTACTS AND LOCATIONS:
Overall Officials: Pebbles Fagan, PhD, MPH, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
To facilitate data use, the research projects will use standard processing and documentation protocols adopted by the Inter-university Consortium for Political and Social Research (ICPSR) for data formats and dictionaries as well as for variable names, descriptions, and labels. We will share all variable de-identified data following the publication of our final results.
Supporting Information: Study Protocol
Time Frame: The data will be made available approximately 1 year after the completion of the study, which is approximately when the final results will be published. ICPSR stores data indefinitely.
Access Criteria: The data are publicly available via ICPSR.